CLINICAL TRIAL: NCT03799133
Title: Safety and Efficacy of the Gastric Reactance (XL) in the Prediction of Morbimortality in Patients Post-operated of Elective Cardiac Surgery
Brief Title: Safety and Efficacy of the Gastric Reactance (XL) in Patients Post-operated of Elective Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Critical Perfusion Inc. (Industry)
Collaborators: Instituto Nacional de Cardiologia Ignacio Chavez (Other); National Council of Science and Technology, Mexico (Other); Gerbera Capital (Other); Alandra Medical SAPI de CV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ISM_VC_01_17; 17-1025 (Other: Instituto Nacional de Cardiología Ignacio Chávez)
Record Dates: First submitted 2018-12-20; First posted 2019-01-10 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Cardiac Failure; Ventricular Dysfunction; Valvular Heart Disease
Keywords: gastric reactance; elective cardiac surgery; morbimortality; APACHE II; STS; SOFA; EUROSCORE II
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction; Heart Valve Diseases

STUDY DESIGN:
Intervention Model Description: Eligible patients will be placed the Florence catheter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Florence device (Experimental): Patients with the Florence catheter placed and connected to the Florence monitor to measure XL trend.
  Interventions: Device: Florence device

INTERVENTIONS:
Device: Florence device — The Florence catheter will be placed at the beginning of the surgery and up to 72 hours in ICU.
  Other Names: ISMO; Gastric Impedance Spectrometer System

SUMMARY:
Evaluate the safety and effectiveness of the XL trend measured by Florence (Critical Perfusion Inc, Palo Alto, California) in the prediction of morbimortality of Mexican patients post-operated of elective cardiovascular surgery.

Hypothesis: 1. The gastric reactance measurement (XL) correlates with the morbimortality (postoperatory shock, excessive bleeding, vasoplegic syndrome and death) and with the risk predictors (APACHE II, STS, SOFA, and EUROSCORE II) with patients post-operated of elective cardiac surgery. 2. It is possible to identify the cut-off point of the values of the gastric reactance (XL) as a predictive tool of morbimortality in patients post-operated of elective cardiac surgery. 3. The gastric reactance (XL) is a safe measurement to patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
A maximum of 35 patients with age greater or equal to 18 years with elective surgery (valvular surgery, revascularization, or a combination of both) that comply with the inclusion/exclusion criteria of this protocol will be enrolled.

Investigational device: Florence (Gastric Impedance Spectrometer System or ISMO). Comparative with Risk scales SOFA, APACHE II, STS, Euroscore II, hemodynamic variables, lactate and mixed venous saturation.

The Florence catheter will be placed at the beginning of the surgery and up to 72 hours in ICU.

ELIGIBILITY:
Inclusion Criteria:

* Women and men within an age equal or greater than 18 years old.
* Subjects scheduled to an elective cardiac surgery for valvular surgery, revascularization or a combination of both.
* Subjects compliant with the indication to be placed a floating pulmonary artery catheter.
* Marks results previous to surgery: STS mortality risk equal or greater than 6% of the day before or Euro Score II with a mortality risk equal or greater than 6% or left ventricle ejection fraction (LVEF/FEVI) less than 45% (patients with cardiac failure or right ventricle dysfunction or a combination of both), tricuspid annular plane systolic excursion (TAPSE) less than 17 mm, peak systolic velocity of tricuspid lateral ring measured by Tissue Doppler (LVOT/TSVI) less than 0.1 m/s; patient with elective surgery of: aortic and mitral valve replacement or aortic and mitral valve replacement + tricuspid valve plasty or aortic valve replacement + mitral valve plasty or mitral valve replacement + tricuspid valve plasty or aortic, mitral and tricuspid valve replacement or aortic valve replacement + tricuspid valve plasty or double valve replacement (any combination) + revascularization or aortic valve replacement + revascularization + mitral valve plasty.
* Subject is not enrolled in another investigational protocol.
* Informed consent has been signed of acceptance by the subject before study procedures.
* Subject in sinus rhythm before surgery.

Exclusion Criteria:

* Subjects with records of recent digestive tube bleeding (last 30 days).
* Paraplegic or hemiplegic subjects.
* Subjects with congenital background (interauricular communication, ventricular atrial channel, coarctation of the aorta, persistent arterial duct, pulmonary stenosis, ventricular septal defect, tetralogy of fallot, total or partial anomalous pulmonary venous drainage, transposition of the great vessels, tricuspid atresia, arterial trunk, etc).
* Maxillofacial malformation.
* Catheter placement failure.
* Known pregnancy or discovered pregnancy after admission (before surgery).
* Woman in breastfeeding period.
* Subjects not compliant with clinical indication of nasogastric catheter placement or contraindicated to place a nasogastric catheter.
* Subjects with an implanted pacemaker or permanent defibrillator.
* Medication supply that impedes contact between Florence catheter and the gastric mucosa (barrier effect) like sucralfate, aluminum hydroxide, bismuth subsalicylate, magaldrate, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2019-12-28 (Actual)

PRIMARY OUTCOMES:
Correlation between gastric reactance (XL) and morbimortality and risk predictors | 72 hours
  Multivariate analysis to observe variability between different events according to data distribution to determine how is affecting the risk scales, hemodynamic variables, lactate and mixed venous oxygen saturation, morbidity and mortality with central gastric reactance (XL).
Sensibility and specificity of the collected variables | 72 hours
  ROC curves will be calculated to determine sensibility and specificity of the variables.
Adverse events tracing with the use of Florence catheter | 30 days
  Serious Adverse Device Effects and Adverse Events assessment to evaluate device safety.

SECONDARY OUTCOMES:
Correlations between XL measurements and medication | 72 hours
  Multivariate analysis to observe variability between different events according to data distribution to determine how is affecting XL with amines, proton-pump inhibitors, and anesthesia medications.
Correlations between laboratory parameters and XL | 72 hours
  Multivariate analysis to observe variability between different events according to data distribution to determine how is affecting XL with laboratory parameters.
Usability of Florence device in a real environment. | 72 hours
  Questionnaire for the nurse and/or the physician regarding the use of Florence device at the Operating Room and Intensive Care Unit.

CONTACTS AND LOCATIONS:
Overall Officials: Rolando J. Álvarez Álvarez, MD, Principal Investigator — Instituto Nacional de Cardiologia Ignacio Chavez; Montserrat Godínez, MSc, Study Director — Alandra Medical SAPI de CV
Locations (1):
- Instituto Nacional de Cardiología Ignacio Chávez, Tlalpan, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- See also: WHO Cardiovascular illness; 2015 — http://www.who.int/mediacentre/factsheets/fs317/es/
- See also: Arias AS, Serrano MEB, Altamirano BD, Ortega MG, Gonzalez GG. Cardiovascular illness: first cause of morbility in a third level hospital. Cardiology Mexican Journal; 2016 — http://www.medigraphic.com/pdfs/cardio/h-2016/hs163a.pdf
- See also: Mittal R, Coopersmith CM. Redefining the gut as the motor of critical illness. Trends in molecular medicine. 2014 Apr;20:214-223 — http://www.ncbi.nlm.nih.gov/pubmed/24055446
- See also: Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, et al. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. Critical care medicine. 2013 Feb;41:580-637 — http://www.ncbi.nlm.nih.gov/pubmed/23361625
- See also: Antonelli M, Levy M, Andrews PJD, Chastre J, Hudson LD, Manthous C, et al. Hemodynamic monitoring in shock and implications for management. International Consensus Conference, Paris, France, 27-28 April 2006. Intensive care medicine. 2007 Apr;33:575-590 — https://www.ncbi.nlm.nih.gov/pubmed/17285286
- See also: Nieminen MS, Boehm M, Cowie MR, Drexler H, Filippatos GS, Jondeau G, et al. Executive summary of the guidelines on the diagnosis and treatment of acute heart failure: the Task Force on Acute Heart Failure of the European Society of Cardiology. — https://www.ncbi.nlm.nih.gov/pubmed/15681577
- See also: McMurray JJV, Adamopoulos S, Anker SD, Auricchio A, Boehm M, Dickstein K, et al. ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure2012 — https://www.ncbi.nlm.nih.gov/pubmed/22611136
- See also: Angus DC, Linde-Zwirble WT, Lidicker J, Clermont G, Carcillo J, Pinsky MR. Epidemiology of severe sepsis in the United States: analysis of incidence, outcome, and associated costs of care. Critical care medicine. 2001 Jul;29:1303-1310 — https://www.ncbi.nlm.nih.gov/pubmed/11445675
- See also: Brun-Buisson C, Meshaka P, Pinton P, Vallet B, Group ES. EPISEPSIS: a reappraisal of the epidemiology and outcome of severe sepsis in French intensive care units. Intensive care medicine. 2004 Apr;30:580-588 — https://www.ncbi.nlm.nih.gov/pubmed/14997295
- See also: Engel C, Brunkhorst FM, Bone HG, Brunkhorst R, Gerlach H, Grond S, et al. Epidemiology of sepsis in Germany: results from a national prospective multicenter study. Intensive care medicine. 2007 Apr;33:606-618 — https://www.ncbi.nlm.nih.gov/pubmed/17323051
- See also: Esteban A, Frutos-Vivar F, Ferguson ND, Penuelas O, Lorente JA, Gordo F, et al. Sepsis incidence and outcome: contrasting the intensive care unit with the hospital ward. Critical care medicine. 2007 May;35:1284-1289 — https://www.ncbi.nlm.nih.gov/pubmed/17414725
- See also: Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, et al.. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3); 2016 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4968574/
- See also: Babaev A, Frederick PD, Pasta DJ, Every N, Sichrovsky T, Hochman JS, et al. Trends in management and outcomes of patients with acute myocardial infarction complicated by cardiogenic shock. JAMA. 2005 Jul;294:448-454 — https://www.ncbi.nlm.nih.gov/pubmed/16046651
- See also: Steg PG, Goldberg RJ, Gore JM, Fox KAA, Eagle KA, Flather MD, et al. Baseline characteristics, management practices, and in-hospital outcomes of patients hospitalized with acute coronary syndromes in the Global Registry of Acute Coronary Events (GRACE). — https://www.ncbi.nlm.nih.gov/pubmed/12161222
- See also: Koek HL, Kardaun JWPF, Gevers E, de Bruin A, Reitsma JB, Grobbee DE, et al. Acute myocardial infarction incidence and hospital mortality: routinely collected national data versus linkage of national registers. European Journal of Epidemiology. 2007 — https://www.ncbi.nlm.nih.gov/pubmed/17828438
- See also: Roger VL, Jacobsen SJ, Weston SA, Goraya TY, Killian J, Reeder GS, et al. Trends in the incidence and survival of patients with hospitalized myocardial infarction, Olmsted County, Minnesota, 1979 to 1994. Annals of internal medicine. 2002 Mar;136:341-348 — https://www.ncbi.nlm.nih.gov/pubmed/11874305
- See also: Geppert A, Steiner A, Zorn G, Delle-Karth G, Koreny M, Haumer M, et al. Multiple organ failure in patients with cardiogenic shock is associated with high plasma levels of interleukin-6. Critical care medicine. 2002 Sep;30:1987-1994 — https://www.ncbi.nlm.nih.gov/pubmed/12352031
- See also: Hamilton MA, Cecconi M, Rhodes A. A systematic review and meta-analysis on the use of preemptive hemodynamic intervention to improve postoperative outcomes in moderate and high-risk surgical patients. Anesthesia and analgesia. 2011 Jun;112:1392-1402 — https://www.ncbi.nlm.nih.gov/pubmed/20966436
- See also: Helander HF, Fändriks L. Surface area of the digestive tract - revisited. Scandinavian journal of gastroenterology. 2014 Jun;49:681-689 — https://www.ncbi.nlm.nih.gov/pubmed/24694282
- See also: Thome JJC, Yudanin N, Ohmura Y, Kubota M, Grinshpun B, Sathaliyawala T, et al. Spatial map of human T cell compartmentalization and maintenance over decades of life. Cell. 2014 Nov; 159:814-828 — https://www.ncbi.nlm.nih.gov/pubmed/25417158
- See also: Reintam B, Poeze M, Malbrain ML, Björck M, Oudemans-van Straaten H. Starkopf J, et al. Gastrointestinal symptoms during the first week of intensive care are associated with poor outcome: a prospective multicentre study. Intensive Care Medicine. 2013 — https://www.ncbi.nlm.nih.gov/pubmed/23370829
- See also: Clark JA, Coopersmith CM. Intestinal crosstalk: a new paradigm for understanding the gut as the "motor" of critical illness. Shock (Augusta, Ga). 2007 Oct; 28:384-393 — https://www.ncbi.nlm.nih.gov/pubmed/17577136
- See also: Klingensmith NJ, Coopersmith CM. The Gut as the Motor of Multiple Organ Dysfunction in Critical Illness; 2016 — https://www.ncbi.nlm.nih.gov/pubmed/27016162
- See also: van Haren FMP, Sleigh JW, Pickkers P, Van der Hoeven JG. Gastrointestinal perfusion in septic shock. Anaesth Intensive Care. 2007 Oct;35(5):679-694 — https://www.ncbi.nlm.nih.gov/pubmed/17933153
- See also: McAdams ET, Jossinet J. Tissue impedance: a historical overview. Physiol Meas. 1995 Aug;16(3 Suppl A):A1-13. Historical Article Journal Article — https://www.ncbi.nlm.nih.gov/pubmed/8528108
- See also: Ivorra A. Bioimpedance monitoring for physicians: an overview; 2003 — http://citeseerx.ist.psu.edu/viewdoc/download?doi=10.1.1.516.4685&rep=rep1&type=pdf
- See also: Kim DW. Detection of physiological events by impedance. Yonsei Med J. 1989;30(1):1-11 — https://www.ncbi.nlm.nih.gov/pubmed/2662632
- See also: Grimnes S, Martinsen OG. Comments on "Algorithm for Tissue Ischemia Estimation Based on Electrical Impedance Spectroscopy". IEEE Transactions on Biomedical Engineering. 2007 Feb;54(2):344-344 — https://ieeexplore.ieee.org/document/4067112
- See also: Rigaud B, Morucci JP, Chauveau N. Bioelectrical impedance techniques in medicine. Part I: Bioimpedance measurement. Second section: impedance spectrometry. Crit Rev Biomed Eng. 1996;24(4-6):257-351 — https://www.ncbi.nlm.nih.gov/pubmed/9196884
- See also: Kun S, Peura RA. Tissue ischemia detection using impedance spectroscopy. In: Engineering in Medicine and Biology Society, 1994. Engineering Advances: New Opportunities for Biomedical Engineers. Proceedings of the 16th Annual International Conference — https://ieeexplore.ieee.org/document/415187
- See also: Ristic B, Kun S, Peura RA. Muscle tissue ischemia monitoring using impedance spectroscopy: quantitative results of animal studies. In: Engineering in Medicine and Biology Society, 1997. Proceedings of the 19th Annual International Conference of the IEEE. — https://ieeexplore.ieee.org/document/758768
- See also: Ivorra A, Genesca M, Sola A, Palacios L, Villa R, Hotter G, et al. Bioimpedance dispersion width as a parameter to monitor living tissues. Physiol Meas. 2005 Apr;26(2):S165-73. Comparative Study Journal Article Research Support, Non-U.S. Gov't — https://www.ncbi.nlm.nih.gov/pubmed/15798229
- See also: Foster KR, Schwan HP. Dielectric properties of tissues and biological materials: a critical review. Critical reviews in biomedical engineering. 1989;17:25-104 — https://www.ncbi.nlm.nih.gov/pubmed/2651001
- See also: Rackow EC, O'Neil P, Astiz ME, Carpati CM. Sublingual capnometry and indexes of tissue perfusion in patients with circulatory failure. Chest. 2001 Nov;120:1633-1638 — https://www.ncbi.nlm.nih.gov/pubmed/11713146
- See also: Rigaud B, Hamzaoui L, Chauveau N, Granie M, Scotto Di Rinaldi JP, Morucci JP. Tissue characterization by impedance: a multifrequency approach. Physiol Meas. 1994 May;15 Suppl 2a:A13-20 — https://www.ncbi.nlm.nih.gov/pubmed/8087035
- See also: Sullivan PG, Wallach JD, Ioannidis JPA. Meta-Analysis Comparing Established Risk Prediction Models (EuroSCORE II, STS Score, and ACEF Score) for Perioperative Mortality During Cardiac Surgery. The American journal of cardiology. 2016 Nov;118:1574-1582 — https://www.ncbi.nlm.nih.gov/pubmed/27687052
- See also: Nashef SAM, Roques F, Sharples LD, Nilsson J, Smith C, Goldstone AR, et al. EuroSCORE II. European journal of cardio-thoracic surgery : official journal of the European Association for Cardio-thoracic Surgery. 2012 Apr;41:734-44; discussion 744-5 — https://www.ncbi.nlm.nih.gov/pubmed/22378855
- See also: A GVO. EuroSCORE II: Como se usa en la practica actual. Revista Mexicana de Cardiologia. 2014 03;25:50 - 51 — http://www.scielo.org.mx/scielo.php?script=sci_arttext&pid=S0188-21982014000100010&nrm=iso
- See also: Vincent JL, de Mendonca A, Cantraine F, Moreno R, Takala J, Suter PM, et al. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working group on "sepsis-related — https://www.ncbi.nlm.nih.gov/pubmed/9824069
- See also: Moreno R, Vincent JL, Matos R, Mendoca A, Cantraine F, Thijs L, et al. The use of maximum SOFA score to quantify organ dysfunction/failure in intensive care. Results of a prospective, multicentre study. Working Group on Sepsis related Problems — https://www.ncbi.nlm.nih.gov/pubmed/10470572
- See also: de Mendonca A, Vincent JL, Suter PM, Moreno R, Dearden NM, Antonelli M, et al. Acute renal failure in the ICU: risk factors and outcome evaluated by the SOFA score. Intensive care medicine. 2000 Jul;26:915-921 — https://www.ncbi.nlm.nih.gov/pubmed/10990106
- See also: Ferreira FL, Bota DP, Bross A, Melot C, Vincent JL. Serial evaluation of the SOFA score to predict outcome in critically ill patients. JAMA. 2001 Oct;286:1754-1758 — https://www.ncbi.nlm.nih.gov/pubmed/11594901
- See also: Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Critical care medicine. 1985 Oct;13:818-829 — https://www.ncbi.nlm.nih.gov/pubmed/3928249
- See also: NIH. Consensus Development Conference on critical care medicine. Critical care medicine. 1983 Jun;11:466-469 — https://www.ncbi.nlm.nih.gov/pubmed/6851607
- See also: Cullen DJ. Results and costs of intensive care. Anesthesiology. 1977 Aug;47:203-216 — http://anesthesiology.pubs.asahq.org/article.aspx?articleid=1960390
- See also: Chalfin DB, Fein AM. Critical care medicine in managed competition and a managed care environment. New horizons (Baltimore, Md). 1994 Aug;2:275-282 — https://www.ncbi.nlm.nih.gov/pubmed/8087584
- See also: O'Brien SM, Shahian DM, Filardo G, Ferraris VA, Haan CK, Rich JB, et al. The Society of Thoracic Surgeons 2008 cardiac surgery risk models: part 2-isolated valve surgery. The Annals of thoracic surgery. 2009 Jul;88:S23-S42 — https://www.ncbi.nlm.nih.gov/pubmed/19559823
- See also: Shahian DM, O'Brien SM, Filardo G, Ferraris VA, Haan CK, Rich JB, et al. The Society of Thoracic Surgeons 2008 cardiac surgery risk models: part 1-coronary artery bypass grafting surgery. The Annals of thoracic surgery. 2009 Jul;88:S2-22 — https://www.ncbi.nlm.nih.gov/pubmed/19559822
- See also: Shahian DM, O'Brien SM, Filardo G, Ferraris VA, Haan CK, Rich JB, et al. The Society of Thoracic Surgeons 2008 cardiac surgery risk models: part 3-valve plus coronary artery bypass grafting surgery. The Annals of thoracic surgery. 2009 Jul;88:S43-S62 — https://www.ncbi.nlm.nih.gov/pubmed/19559824
- See also: Rankin JS, He X, O'Brien SM, Jacobs JP, Welke KF, Filardo G, et al. The Society of Thoracic Surgeons risk model for operative mortality after multiple valve surgery. The Annals of thoracic surgery. 2013 Apr;95:1484-1490 — https://www.ncbi.nlm.nih.gov/pubmed/23522221